CLINICAL TRIAL: NCT05682456
Title: High-fat Challenge Induced Trained Innate Immunity
Brief Title: High-fat Challenge Induced Trained Innate Immunity (SHAKE Study)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Radboud University Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: 107808; NTR7612 (Registry Identifier: Netherlands Trial Register)
Record Dates: First submitted 2022-12-16; First posted 2023-01-12 (Actual); Last update posted 2023-01-12 (Actual); Status verified 2022-12

CONDITIONS: Cardiovascular Diseases
MeSH Terms: conditions — Cardiovascular Diseases

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- High-fat shake (Experimental)
  Interventions: Dietary Supplement: High-fat shake
- Reference shake (Active Comparator)
  Interventions: Dietary Supplement: Reference shake

INTERVENTIONS:
Dietary Supplement: High-fat shake — The high-fat shake consisted of 53% (w/v) fresh cream, 3% (w/v) sugar and 44% (w/v) water
  Arms: High-fat shake
Dietary Supplement: Reference shake — The reference shake consisted of 43% (w/v) full cream milk, 48% (w/v) full cream yoghurt, 4% (w/v) lemonade, 4% (w/v) fantomalt (Nutricia B.V., the Netherlands) and 1% (w/v) wheat fiber
  Arms: Reference shake

SUMMARY:
The goal of this randomized controlled cross-over trial is to investigate whether a single high-fat challenge can induce trained innate immunity in healthy volunteers. The main question it aims to answer is: Can a single high-fat challenge induce a persistent pro-inflammatory and pro-atherogenic monocyte phenotype, as detected by an augmented cytokine production capacity? To study this, participants will receive an oral high-fat and reference shake in a cross-over design and blood will be drawn before and at 1, 2, 4, 6, 24, and 72 hours after the shakes.

DETAILED DESCRIPTION:
Rationale: Atherosclerosis is characterized by a persistent inflammation of the arterial wall.

Monocyte-derived macrophages are the most abundant immune cells in atherosclerotic plaques. It has recently been shown that not only immune cells of the adaptive immune system, but innate immune cells as well are able to adopt a long-term pro-inflammatory phenotype upon stimulation. This nonspecific memory of innate immune cells is mediated by epigenetic and metabolic reprogramming and is termed "trained innate immunity." Previous findings from our lab have shown that not only bacterial components such as LPS, but also pro-atherogenic particles such as oxidized LDL can induce trained immunity in monocytes. Interestingly, this memory-effect of trained immunity indicates that even temporary triggers could induce the persistent inflammation in atherosclerosis.

Triglyceride-rich lipoproteins (TRL) have been identified as an important independent risk factor for atherosclerosis. Moreover, elevated plasma levels of these lipoproteins are associated with increased pro-inflammatory markers. TRLs, however, are characterized by alternating plasma levels, with brief elevations following (fat containing) meals. Notably, a high-fat meal not only contributes to the transient increase of TRL plasma levels, but also induces a brief elevation in LPS levels by briefly increasing the permeability of the gut.

We now aim to investigate whether a single high-fat meal can induce trained innate immunity, since this concept might explain how brief postprandial effects can translate into a long-term pro-inflammatory and pro-atherogenic monocyte phenotype.

Objective: The primary objective is to determine whether a high-fat meal can induce a persistent pro-inflammatory monocyte phenotype, characterized by an increased cytokine production capacity upon ex vivo stimulation. Secondary objectives are metabolic and epigenetic reprogramming of monocytes at these time points as well as the capacity of serum, isolated before and 1-6h after an oral fat load, to induce an increased cytokine production in healthy human monocytes.

Study design: Randomized cross-over high-fat challenge intervention study.

Study population: Healthy human volunteers, aged between 18 and 40 years.

Intervention: A single high-fat challenge (milkshake containing 95g of fat) and 'control' shake (comparable to an average breakfast).

Main study parameters/endpoints: Blood will be drawn at t=0h (before) and at t=1h, t=2h, t=4h, t=6h, t=24 and t=72h after an oral fat load and at the same time points after a 'control' shake. The primary endpoint is the monocyte TNFα production upon ex vivo stimulation with LPS at the 72h time point. Additional secondary endpoints are the production of other cytokines and chemokines upon ex vivo stimulation at t=0h, t=4h, t=24h and t=72h, the monocytes' inflammatory phenotype as assessed by flowcytometry analysis and serum induced persistent cytokine production capacity.

ELIGIBILITY:
Inclusion Criteria:

* LDL cholesterol < 3.5 mmol/l, fasting triglycerides < 2 mmol/l
* No previous cardiovascular events

Exclusion Criteria:

* Smoking within the year before study entry
* Diagnosed with any long-term medical condition that can interfere with the study (i.e.

gallbladder disease, renal failure, cardiovascular disease, diabetes, rheumatoid arthritis etc.)

* Medication (with the exception of oral contraceptives) or supplement use (i.e. omega3)
* BMI < 18 or > 27 kg/m2
* Previous vaccination within 3 months prior to study entry
* Current infection or clinically significant infections within 1 month before study entry (defined as fever > 38.5°C)
* Allergic to cow milk/dairy products
* Pregnancy/lactation
* Abuse of drugs or alcohol
* Vegetarian diet

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 16 (Actual)
Dates: Start 2019-05-06 (Actual); Primary Completion 2020-01-09 (Actual); Study Completion 2021-10-15 (Actual)

PRIMARY OUTCOMES:
Monocyte TNFα production upon ex vivo stimulation with LPS | 72 hours

SECONDARY OUTCOMES:
The monocyte production of TNFa, IL-6, IL-1beta, IL-10 upon ex vivo stimulation with LPS, Pam3Cys or Candida Albicans. | 0 hour, 4 hours, 24 hours and 72 hours
The monocyte's inflammatory phenotype as assessed by flowcytometry analysis (i.e. membrane expression of markers including but not limited to CD14, CD16, CD11b, CCR2) | 0 hour, 4 hours, 24 hours and 72 hours
Postprandial serum-induced TNFa and IL-6 production of healthy human monocytes upon stimulation with LPS or Pam3Cys 6 days later. | 0 hour, 2 hours, 4 hours , 6 hours
  Serum isolated before and after consumption of a high-fat meal is used in in vitro studies. In these studies isolated monocytes of healthy human donors are exposed to pooled fasting (t=0h) or fed serum (t=2h, 4h, or 6h) obtained from the study participants. The TNFa and IL-6 production of these cells is measured after stimulation with LPS and Pam3Cys 6 days later. Subsequently, it is studied whether a possible increase in TNFa or IL-6 production can be prevented by co-incubation with pharmacological inhibitors (e.g. TLR4 antagonists/inhibitors)
Plasma triglyceride, glucose, free fatty acid and insulin concentrations | 0 hour, 1 hour, 2 hours, 4 hours , 6 hours
  The baseline (t=0h) and postprandial concentrations (at t=1h, 2h, 4h and 6h) of circulating triglycerides, glucose, free fatty acids and insulin are measured in the study participants after consumption of both the high-fat and control shake.

CONTACTS AND LOCATIONS:
Overall Officials: Niels Riksen, MD, PhD, Principal Investigator — Vascular Internal Medicine, Radboudumc
Locations (1):
- Radboudumc, Nijmegen, Gelderland, Netherlands

IPD SHARING:
Plan to Share IPD: Undecided